CLINICAL TRIAL: NCT00702130
Title: The Effect of Pravastatin on the Incidence and in the Natural Course of Ventilatory Associated Pneumonia in the Intensive Care Unit Patients
Brief Title: Pravastatin and Ventilatory Associated Pneumonia
Acronym: EPRAVAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Efstratios Manoulakas, Ph, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 310UT
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): this arm will receive Pravastatin 40 mg per os daily
  Interventions: Drug: Pravastatin
- 1 (No Intervention)

INTERVENTIONS:
Drug: Pravastatin — pravastatin 40mg per os once daily
  Arms: A

SUMMARY:
Statins present anti-inflammatory and immunomodulatory effects. They may modify the regulation of cytokines, (released from the cellular damage) and may reduce the production of C-reactive protein levels. It has been hypothesized that these pleiotropic characteristic of statins might be useful in the management of various diseases, including pneumonia. Indeed, a recent study showed that statin treatment is associated with reduced risk of pneumonia in diabetic patients. However, the relationship between statins and reduced risk of pneumonia is not consistent . In addition there is no prospective study to investigate the role of statins in severe forms of pneumonia such as the VAP.

On this base the investigators aim to study prospectively the effect of statins on the outcome of patients with VAP in the ICU settings. The investigators therefore contacted a double open label randomized trial to investigate whether the use of pravastatin reduces the incidence of Ventilator Associated Pneumonia in the ICU and whether it is related with favorable outcome of patients with Ventilator Associated Pneumonia.

DETAILED DESCRIPTION:
INTRODUCTION

The pneumonia in the intensive care unit (I.C.U.) constitutes the most frequent infection and is most often associated with the application of the mechanical ventilation. VAP (Ventilator - Associated Pneumonia) is defined as the nosocomial pneumonia in a patient on mechanical ventilatory support (by endotracheal tube or tracheostomy) for more than 48 hours. The risk for such complication is proportionally increased with the duration of hospitalization. The symptoms include the appearance of pulmonary infiltrate, fever, leukocytosis and purulent tracheobronchial secretions although this symptomatology is not always present. VAP is usually caused by several nosocomial species, such as Acinetobacter baumanni (the most often), Pseudomonas aeruginosa, Klebsiella pneumoniae.

VAP is frequently complicated with the entry of bacteria in the circulation of blood resulting in bacteremia and sepsis. In this respect, this disorder is associated with substantial morbidity and devastating costs of hospitalization. Notably, the cost of one episode of VAP is estimated in 57000 $ per occurrence.

On this basis, several strategies have been implicated to minimize the risk of VAP and to manage effectively the disease (5-12). Among these, antinflammatory treatment has been used in the past to influence the course of and to alter favorably the outcome of VAP (13).

Statins (HMG-CoA-reductase inhibitors), are drugs that regulates the speed of composition of cholesterol suspending the composition of cholesterol in very precocious stage. Recent studies have brought in the surface new attributes of statins. Statins present anti-inflammatory and immunomodulatory effects. They may modify the regulation of cytokines, (released from the cellular damage) and they may reduce the production of C-reactive protein levels (14-19). It has been hypothesized that these pleiotropic characteristic of statins might be useful in the management of various diseases (20), including pneumonia. Indeed, a recent study showed that statin treatment is associated with reduced risk of pneumonia in diabetic patients (18). However, the relationship between statins and reduced risk of pneumonia is not consistent (19). In addition there is no prospective study to investigate the role of statins in severe forms of pneumonia such as the VAP. We therefore contacted a double open label randomized trial to investigate whether the use of pravastatin reduces the incidence of Ventilator Associated Pneumonia in the ICU and whether it is related with favorable outcome of patients with Ventilator Associated Pneumonia.

MATERIALS AND METHODS

Study population and protocol The present is a prospective randomized open label controlled trial. The study will take place in the intensive care (ICU)of the University Hospital of Larissa and the General Hospital of Larissa in Greece.

Consecutive sampling will be used to recruit patients hospitalized in the ICU department between June of 2008 and August of 2009. The patients will be randomized to receive pravastatin sodium 40 mg (subjects) or not (controls). The trial medication will be commenced within 24 hours of ICU admission (Day 0). The treatment group will receive pravastatin for up to 30 days.

Authorization has been given from the Scientific Council and the Ethical Committee of our Hospital.

Diagnosis of VAP will be based on the following definition (1): the appearance of a new and persistent pulmonary infiltrate on chest radiography, fever (>38.2ºC), leukocytosis or leukopenia (>12000/mm³ or <4000/mm³ respectively), purulent tracheobronchial secretions and microbiological documentation by bronchial aspirated or BAL.

Clinical assessment and microbiology Prerandomization baseline assessment will include evaluation of demographic data, medical history, radiography of thorax, blood leukocyte count, PaO2/FiO2, maximum body temperature of the day, CRP levels, the APACHE score in the entrance in ICU, the SOFA score, Murray score and the serum amyloid alpha levels. Measurements of the above parameters will take place at the baseline (Day 0), at the 5th, 10th, 20th of admission, at the day of VAP diagnosis and at the 3rd, 5th, 10th of VAP and at the day of discharge from the ICU.

Microbiology To determine bacterial species responsible for VAP, bronchial secretions or BAL will be sampled at the baseline (Day 0), at the 5th, 10th, 20th of admission, at the day of VAP diagnosis and at the 3rd, 5th, 10th of VAP and at the day of discharge from the ICU. Samples will be also collected at any other day if the attending physician finds it clinically significant according to established protocol (22). Microbiology assessment will include identification of the responsible agent (Gram and culture) in bronchial secretions and BAL (50cc NaCl 0.9%) and assessment of antibiotic resistance. Accordingly bacterial species will be categorized as sensitive to colistin or not (1-3).

VAP Management and monitoring Treatment of VAP will be based on the attending physician decision according to guidelines. All relevant diagnostic and therapeutic decisions will be discussed in a daily multidisciplinary ICU meeting (5-12).

Clinical follow up of the patients will be continued for up to 6 months from the initiation of the study to document late adverse events related to the study.

Statistical Analysis All analysis will be performed on an intention-to-treat basis, and probability values will be 2-sided. Data will be presented as mean +/- SD and 95% CI. Analysis will be performed using statistical software, SISS 15 for Windows. Data will be compared between the pravastatin and the control groups. Pre- and post- randomization characteristics will be compared using the χ² test (the Fisher exact test will be used when any number off the cell will be <5) and the t test. Stepwise multiple logistic or linear regression analysis will be applied to determine the factors that might the factors that might be considered independent predictors of unfavorable outcome and scores, whereas a significance level of 0.05 will be chosen for variable entry into the model. The odds ratio (OR) and linear coefficient will be calculated and presented with 95% CI. P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Presence in Intensive Care Unit

Exclusion Criteria:

* Pregnancy,
* Pneumonia, previous use of statins,
* Contraindications to statin use (liver dysfunction, SGOT/SGPT > 100 U/L),
* Increased CPK (over 3 times the upper limit), (for non trauma patients) on admission,
* Increase of CPK (over 5 times the upper limit) during hospitalization,
* Use of substances that contraindicates simultaneous use of statins (macrolides, cyclosporine, antipyrin, cholestyramine, gemfibrosil, warfarin),
* Malabsorption syndrome (over the first 48 hours).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization in the Intensive Care Unit, morbidity in the Intensive Care Unit | 1 year

SECONDARY OUTCOMES:
Severity of Ventilator Associated Pneumonia | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - General Hospital Larissa, Larissa, Thessaly
  - Zakynthinos E. Dir-University Hospital Larisa, Mezourlo / Larissa